CLINICAL TRIAL: NCT03873727
Title: Evaluation of Immunological Response Following a Revaccination With PPS23 Boosted or Not by PCV13 in Splenectomised Patients
Brief Title: Revaccination With PPS23 Boosted or Not by PCV13 in Splenectomised Patients.
Acronym: SPLENEVAC-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: EUCLID Clinical Trial Platform (Other); Recherche Clinique Paris Descartes Necker Cochin Sainte Anne (Other); CIC 1417 Cochin-Pasteur (Other); I-REIVAC Innovative Clinical Research Network In Vaccinology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P170934J; 2018-003068-29 (EudraCT Number)
Record Dates: First submitted 2019-02-12; First posted 2019-03-13 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Splenectomised Patients
Keywords: Vaccination / Re-vaccination; Asplenic patient; Splenectomy; Pneumococcal infections; immunological response; Pneumovax; Prevenar13
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine; Pneumococcal Vaccines; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevenar13/ Pneumovax (Experimental): Prime-boost strategy combining a single dose of 13-valent pneumococcal conjugate vaccine (Prevenar 13, PCV13) at month 0 (M0) followed by a single dose of 23-valent unconjugated vaccine (Pneumovax, PPS23) at month 12 (M12).
  Interventions: Biological: Prevenar13 (PCV13) and Pneumovax (PPS23); Biological: Blood sample
- Placebo / Pneumovax (Placebo Comparator): Standard strategy combining a single dose of placebo vaccine (Prevenar 13 placebo) at month 0 (M0) followed by a single dose of 23-valent unconjugated vaccine (Pneumovax, PPS23) at month 12 (M12)
  Interventions: Biological: Placebo / Pneumovax (PPS23); Biological: Blood sample

INTERVENTIONS:
Biological: Prevenar13 (PCV13) and Pneumovax (PPS23) — One dose of PCV13 at Month 0 and one dose of PPS23 at Month 12
  Arms: Prevenar13/ Pneumovax
Biological: Placebo / Pneumovax (PPS23) — One dose of Placebo at Month 0 and one dose of PPS23 at Month 12
  Arms: Placebo / Pneumovax
Biological: Blood sample — an additional 5 mL sample of blood at one of the visits, preferably at the first visit, concerning patients included in Parisian centers who did not participate in SPLENEVAC 1 study.

SUMMARY:
This research is a multi-center French randomized and double blind phase IIb clinical trial evaluating 2 revaccination strategies against pneumococcal infections among splenectomised patients. The main objective is to evaluate at M13 the immunological response of 2 pneumococcal revaccination strategies (combined revaccination by a boost dose of PCV13 following 12 months later by PPS23, versus PPS23 alone) in splenectomised adults.

DETAILED DESCRIPTION:
For the prevention of invasive pneumococcal diseases, two polysaccharide vaccines are currently available: a non-conjugate vaccine, Pneumovax® (PPS23), and a conjugate vaccine, Prevenar13® (PCV13), inducing protection against 23 and 13 pneumococcal serotypes, respectively. The PPS23 is considered weakly immunogenic, especially in infants, elderly and immunocompromised patients, while PCV13 is now available for adults. In France, in April 2017, the new recommendations for at risk patients including asplenic patients are to revaccinate by PPS23 at least five years after the previous PPS23. However a phenomenon of vaccine hyporesponsiveness and a risk of immune tolerance to pneumococcus after repeated administrations of PPS23 are described. Large doses of polysaccharide antigens recruit memory and naive B cells, resulting in the production of low and high avidity antibodies, while low doses only stimulate memory B cells, inducing high affinity antibodies. Because of that, Swiss current recommendations are to revaccinate with PCV13 at 5 years the splenectomised patients. The recommendations of revaccination by PPS23 for USA or PCV13 for Switzerland have never been evaluated in clinical trial. Moreover, using combined PCV13/PPS23 could increase serotype coverage. Studying the immune response following combined revaccination by a boost dose of PCV13 following by PPS23 versus PPS23 alone will help to document and improve the vaccine recommendations.

The main objective is to evaluate at M13 the immunological response of 2 pneumococcal revaccination strategies (combined revaccination by a boost dose of PCV13 following 12 months later by PPS23, versus PPS23 alone), in splenectomised adults.

The primary endpoint is the proportion of patients responding to a minimum of 5 of the 9 serotypes analysed (9 serotypes among the 12 common serotypes to both PPS23 and PCV13: 1, 3, 6B, 7F, 9V, 14, 19A, 19F, and 23F) at M13 in each arm. A responder to a serotype is defined as a four-fold increase of the rate of OPA (OpsonoPhagocytic Assay) compared to baseline and titer ≥ LLOQ (Lower Limit of Quantification).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Splenectomised patients.
3. For patients not enrolled in SPLENEVAC clinical trial: presence of Jolly Body at blood smear and spelenectomy confirmation by abdominal ultrasound.
4. Vaccinated according to the schedule of SPLENEVAC clinical trial (PCV13 / PPS23 two months later (until +4 months)), enrolled or not from this study. Vaccination of PPS23 must have been administered 5 years - 6 months/+ 1 year before inclusion.
5. Patients will be followed during the 24 months from the inclusion visit.
6. Patients must give written informed consent prior to any trial procedure.
7. Women of childbearing age must have an effective contraception during the first 13 months of the study.
8. Patients must be covered by social security regimen or equivalent.

Exclusion Criteria:

1. History of pneumococcal revaccination in the last five years.
2. Having received any another vaccines within 4 weeks prior to enrolment or who is planning to receive any vaccine (for example: ZOSTAVAX®) within the first 13 months of the study (excepted seasonal influenza vaccine which is permitted 4 weeks before and after each vaccination visit of the study and then allowed at any time during the study follow up. Furthermore, the vaccination against Sars-CoV-2 is allowed during the study with a minimum interval of 14 days between pneumococcal vaccine and Sars-Cov-2 vaccine injection)
3. History of known allergies to any component of both study vaccines (active substances, excipients or diphtheria toxoid).
4. History of anaphylactic reaction following vaccination.
5. Infusion of immunoglobulins within the three months preceding the inclusion.
6. Any pathology or condition that may impair the immune response, apart from splenectomy: immunosuppressive therapy in progress or in the 6 months prior to inclusion, hematopoietic stem cells allo / autograft, primary immunodeficiency, nephrotic syndrome, progressive neoplasia, evolutive cancer, cirrhosis, known infection to HIV and / or hepatitis B virus (HBV) (HBs Ag +) and / or hepatitis C virus (HCV), taking corticosteroids > 10mg for more than 14 days within the month preceding the inclusion , inhaled corticosteroid and cutaneous topical being allowed.
7. Coagulation disorder contra-indicating intramuscularly injections.
8. Acute respiratory tract infection or severe acute febrile illness or systemic reaction which could represent a significant risk in case of vaccination within the month before inclusion.
9. Pregnancy, breastfeeding or positive pregnancy test up to 13 months after inclusion.
10. History of suspected or documented invasive pneumococcal infection within the year before inclusion.
11. Immunosuppressive factors associated.
12. Enrolment in any other clinical trial during the whole trial period except observational study.
13. Adults under protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity | at Month 13
  Immune response at M13 against minimum of 5 of the 9 serotypes analysed (9 serotypes among the 12 common serotypes to both PPS23 and PCV13: 1, 3, 6B, 7F, 9V, 14, 19A, 19F, and 23F) in each arm.
  A responder to a serotype is defined as a four-fold increase of the rate of OpsonoPhagocytic Assay (OPA) compared to baseline (M0) and titer ≥ Lower Limit of Quantification (LLOQ).

SECONDARY OUTCOMES:
Enzyme-linked immunosorbent assay (ELISA) antibody dosages | Month 0 to Month 24
  ELISA antibody concentration against 9 common serotypes (1, 3, 6B, 7F, 9V, 14, 19A, 19F and 23F), and, the proportion of positive serotypes: serotype is considered positive if the immunoglobulin G (IgG) antibody concentration in ELISA shows a two-fold increase from baseline (M0) in each arm from baseline.
Enzyme-linked immunosorbent assay (ELISA) antibody dosages | Month 0 to Month 24
  ELISA antibody concentration against 9 common serotypes (1, 3, 6B, 7F, 9V, 14, 19A, 19F and 23F), and, the proportion of positive serotypes: serotype is considered positive if the IgG antibody concentration is ≥ 1μg/ml in each arm from baseline.
Enzyme-linked immunosorbent assay (ELISA) antibody dosages | Month 0 to Month 24
  ELISA antibody concentration against 9 common serotypes (1, 3, 6B, 7F, 9V, 14, 19A, 19F and 23F), and, the proportion of positive serotypes: serotype is considered positive if the IgG antibody concentration shows a two-fold increase from baseline (M0) in each arm and IgG ≥ 1μg/ml from baseline.
Titration of OPA - | at Month 0, Month 13 and Month 24
  OPA titers against 9 common serotypes (1, 3, 6B, 7F, 9V, 14, 19A, 19F and 23F) and the proportion of positive serotype: serotype is considered positive if the antibody titer shows a four-fold increase from baseline (M0).
Titration of OPA - | at Month 0, Month 13 and Month 24
  OPA titers against 9 common serotypes (1, 3, 6B, 7F, 9V, 14, 19A, 19F and 23F) and the proportion of positive serotype: serotype is considered positive if the antibody titer ≥ LLOQ.
Titration of OPA - | at Month 0, Month 13 and Month 24
  OPA titers against 9 common serotypes (1, 3, 6B, 7F, 9V, 14, 19A, 19F and 23F) and the proportion of positive serotype: serotype is considered positive if the antibody titer shows a four-fold increase from baseline (M0) and titer ≥ LLOQ.
ELISA antibody dosages | at Month 12, Month 13 and Month 24
  ELISA antibody concentration against 3 uncommon specific serotypes of PPS23 (12F, 10A and15B) and the proportion of positive serotypes: serotype is considered positive if the IgG antibody concentration shows a two-fold increase from baseline (M12) in each arm and IgG ≥ 1 μg/ml
ELISA antibody dosages | at Month 12, Month 13 and Month 24
  ELISA antibody concentration against 3 uncommon specific serotypes of PPS23 (12F, 10A and 15B) and the proportion of positive serotypes: serotype is considered positive if the IgG antibody concentration shows a two-fold increase from baseline (M12) in each arm.
ELISA antibody dosages | at Month 12, Month 13 and Month 24
  ELISA antibody concentration against 3 uncommon specific serotypes of PPS23 (12F, 10A and 15B) and the proportion of positive serotypes: serotype is considered positive if the IgG antibody concentration in ELISA is ≥ 1μg/ml in each arm.
Sustainability and evolution of the immune response | at Month 0 and Month 24
  Measure of ELISA concentration and OPA titers for the 9 PCV13 serotypes in each arm.
ELISA antibody dosages | at Month 3
  ELISA antibody concentration against 9 common specific serotypes (1, 3, 6B, 7F, 9V, 14, 19A, 19F and 23F) and the proportion of positive serotype: serotype is considered positive if the IgG antibody concentration in ELISA and shows a two-fold increase from baseline (M0) in each arm in SPLENEVAC 1
Percentage of patients presenting local or systemic reactions post-immunization | Month0 to Month 24
  Number of subjects with local and systemic reactions following vaccinations (tolerability) in each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, MD,PhD, Principal Investigator — CIC 1417 Clinical Center Investigation - Cochin Hospital, AP-HP; Olivier Lortholary, Md,PhD, Principal Investigator — Service des Maladies Infectieuses et Tropicales, Necker-Enfants malades Hospital, AP-HP; Hélène Coignard-Biehler, MD,PhD, Principal Investigator — COREB - Hospices Civils de Lyon; Marc Michel, MD,PhD, Principal Investigator — Service de médecine interne, Henri Mondor Hospital, APHP; Benjamin Rossi, MD, Principal Investigator — Service de Médecine interne et de Maladies infectieuses, Robert Ballanger Hospital
Locations (1):
- CIC 1417 Cochin-Pasteur - GH Broca-Cochin-Hôtel-Dieu, Paris, France

IPD SHARING:
Plan to Share IPD: No